CLINICAL TRIAL: NCT06855303
Title: Comparison Between the Effects of Two Different Muscle Energy Techniques on Hamstring Flexibility in Patients With Hamstring Tightness Secondary to Knee Osteoarthritis: Randomized Controlled Trial
Brief Title: Muscle Energy Technique and Muscle Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, associate professor, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-2025-585
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-03

CONDITIONS: Hamstring Shortness

STUDY DESIGN:
Intervention Model Description: The study model will include 2 parallel groups of equal number. Each group will receive a different variation of muscle energy technique (MET)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants will be assigned to the groups using permuted block design. The number of blocks will be 4 and 6. The person (not involved in assessment nor treatment) who will be responsible for allocation will give each participant a code number indicating his/her group. only the therapist will be allowed to reveal the code number interpretation to provide the appropriate intervention, while patients, the assessor, and the data analyzer (statistician) will be kept blind throughout the study. regarding the statistician, the raw data will be sent after removal of the group name, which will be replaced by a code letter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Experimental): this arm will receive muscle energy technique using the post isometric relaxation principle
  Interventions: Other: Muscle Energy Teqnique using post isometric relaxation (PIR) principle; Other: Conventional Treatment group
- group 2 (Experimental): this group will recieve muscle energy technique using the receprocal inhibition (RI) principle
  Interventions: Other: Muscle Energy Teqnique using receprocal inhibition (RI) principle; Other: Conventional Treatment group
- group 3 (Active Comparator): This group will receive a 10-minute application of high-frequency TENS. Hot moist pack: The patient will be made to lie in a supine position with the affected knee in slight flexion. A hot moist pack will be applied around the knee for 15 minutes. Ankle pumps, Heel slides, Open chain knee flexion and extension exercises, Straight leg raise, Quad isometrics and Calf stretch. All these exercises were given 10 repetitions x1 set, three days/week.
  Interventions: Other: Conventional Treatment group

INTERVENTIONS:
Other: Muscle Energy Teqnique using post isometric relaxation (PIR) principle — The contralateral leg may be either flexed or may lie straight on the plinth. The affected leg will be flexed at both the hip and knee joints, and then slowly straightened by the therapist until the restriction barrier is identified. The limb will be moved a little away from the restriction barrier and the isometric contraction against resistance is introduced. The patients will be asked to resist the movement with no more than 25% of strength. The contraction will be held for 7-10 seconds followed by complete relaxation of the limb. On exhalation, the knee joint will be straightened (extended) towards its new barrier, and through that barrier a stretch will be applied and maintained for 30 seconds. 3 repetitions
  Arms: group 1
Other: Muscle Energy Teqnique using receprocal inhibition (RI) principle — The supine patient will ask to fully flex the hip and knee on the affected side. The affected leg will then be slowly straightened by the therapist until the restriction barrier is identified. The calf of the affected leg will then be placed on the practitioner's shoulder that stands facing the head of the table on the side of the affected leg. Then the patient will be asked to attempt to straighten the lower leg utilizing the antagonists to hamstrings, employing approximately 20 percent of the strength of the quadriceps. This will be resisted by the practitioner for 5 to 7 seconds. Appropriate breathing instructions will be given. On exhalation, the knee joint will be straightened (extended) towards its new barrier and through that barrier a stretch will be applied and maintained for 30 seconds. 3 repetitions)four repetition
  Arms: group 2
Other: Conventional Treatment group — This group will receive a 10 minutes application of high-frequency TENS. Hot moist pack: The patient will be made to lay in a supine position with the affected knee in slight flexion A hot moist pack will be applied around the knee for 15 minutes. Ankle pumps, Heel slides, Open chain knee flexion and extension exercises, Straight leg raise, Quad isometrics and Calf stretch. All these exercises were given 10 repetitions x1 set, three days/week

SUMMARY:
The current study will compare the effect of using the muscle energy technique in 2 different methods on the hamstring muscle flexibility

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a painful musculoskeletal disease that primarily affects the knee, resulting in the gradual degeneration of articular cartilage. Knee OA commonly affects the elderly population and may cause impairment throughout the world. About 4% of the world's population suffers from osteoarthritis, especially in those who are 50 years of age or older.

Age, trauma, congenital and acquired deformity, metabolic conditions, obesity, muscle weakness or imbalance, an occupation that requires prolonged sitting and knee bending, and female gender are all risk factors linked to the development of Knee OA.

Knee pain, morning stiffness, knee locking, or giving way, crepitus, and functional impairments are the common clinical symptoms of Knee OA.

Initial treatment always begins with conservative modalities and progresses to surgical treatment when conservative treatment fails. There is a variety of conservative techniques available for the treatment of knee OA.

The two main muscles that move the knee joint are the quadriceps and hamstrings, which help the knee joint's ambulatory growth factors move smoothly and precisely.

The hamstring muscles are noted for their tendency to shorten, and knee OA has been linked to decreased hamstring flexibility that can put more strain on the knee joint, reduce range of motion, and walking abnormalities. Furthermore, reduced flexibility can result in patellofemoral syndrome, which can cause pain and restrictions in physical functioning and increase the compressive load on the patellofemoral joint. Patellofemoral syndrome frequently contributes to osteoarthritis.

In general, when muscle is flexible, the body may avoid unnecessary energy expenditure and improve movement accuracy, strength, and coordination to ensure that muscles and joints can move freely. Therefore, increasing hamstring flexibility can aid in relieving symptoms and reducing knee joint pressure in patients with knee OA.

The first-line treatment for all symptomatic knee OA patients includes education and physiotherapy. Among the physiotherapy techniques, muscle energy techniques (MET) like post-isometric relaxation (PIR) and reciprocal inhibition (RI) have become popular due to their efficacy in relaxing and lengthening muscles, reducing pain, and improving overall function in patients with knee OA. Furthermore, MET helps the body drain blood and bodily fluids through the lymphatic or venous pumps, strengthen muscles, and increase the range of motion in joints with limited range of motion.

Numerous studies have demonstrated the benefits of MET in improving function, flexibility, and pain in knee OA patients. For example, MET may be more beneficial than conventional treatments in enhancing knee OA patients' flexibility and functional outcomes, whether used with or without other techniques.

However, few studies have compared the relative effectiveness of various MET approaches in treating knee OA patients' flexibility, pain, and joint mobility problems.

Finally, the majority of research regarding the impact of the MET on hamstring flexibility has brief observation periods involving small samples and low quality, primarily focusing on healthy individuals under the age of 45. Consequently, additional high-quality research should evaluate the efficacy of MET on hamstring flexibility required with larger sample sizes that include older age groups.

Therefore, more research is required to evaluate the impact of different MET on hamstring flexibility in knee OA patients.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically and clinically diagnosed cases of Osteoarthritis knee by a certified Orthopaedic surgeon or Physiotherapist. Patients with Grade 2 or 3. Osteoarthritis knee according to Kellgren - Lawrence classification,
* Between the age group of 40-60 years, including both men and women.
* Hamstring tightness of more than 20 from the active knee extension test (AKET)

Exclusion Criteria:

* Other knee joint pathologies such as Chondromalacia patella, plica syndrome,
* Neurological disorders.
* Patients having lower extremity injury/surgeries in the past 6 months,
* Hip or knee fractures or deformity,

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
The Numeric Pain Rating | From baseline to the end of the treatment at 6 weeks
  The numeric pain rating Scale (NPRS) is the simplest and most commonly used numeric scale to rate the pain from 0 (no pain) to 10 (worst pain). The NPRS will be used for subjective pain measurement that has good test-retest reliability.
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | From baseline to the end of the treatment at 6 months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) will be used to measure symptoms and physical disability, originally developed for people with OA of the hip or knee. It evaluates three dimensions: pain, stiffness, and physical function
Sit and reach test | From baseline to the end of the treatment at 6 weeks
  The Sit and reach test is one of the linear flexibility tests that helps to measure flexibility of the lower back and hamstring muscles.
  equipment required: sit and reach box (or alternatively a ruler can be used, and a step or box).
  procedure: This test involves sitting on the floor with legs stretched out straight ahead. Shoes should be removed. The soles of the feet are placed flat against the box. Both knees should be locked and pressed flat to the floor - the tester may assist by holding them down. With the palms facing downwards, and the hands on top of each other or side by side, the subject reaches forward along the measuring line as far as possible. After some practice reaches, the subject reaches out and holds that position for at least one to two seconds while the distance is recorded.
  Ayala et al. showed acceptable reproducibility measures for the sit and reach test with 8.74% coefficient of variation (CV) and 0.92 intraclass correlation coe

CONTACTS AND LOCATIONS:
Overall Officials: Hisham M Hussein, PhD, Principal Investigator — University of Hail
Locations (1):
- University of Hail, Hail, Ha'il Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
because they will be used in other future studies